CLINICAL TRIAL: NCT01813565
Title: The Efficacy of Additional Intravesical Instillation of Hyaluronic Acid/Chondroitin Sulfate to Transurethral Resection of Bladder Ulcer in Patients With Interstitial Cystitis/Bladder Pain Syndrome.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: No benefit of intravesical instillation of Hyaluronic Acid/Chondroitin Sulfate
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Myung-Soo Choo, Profesor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20130135
Record Dates: First submitted 2013-03-11; First posted 2013-03-19 (Estimated); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Interstitial Cystitis
MeSH Terms: conditions — Cystitis, Interstitial | interventions — Hyaluronan Receptors; chondroitin sulfate, sodium hyaluronate drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Additional instillation of hyaluronic acid/chondroitin sulfate (Experimental): Transurethral resection of bladder ulcer + instillation of hyaluronic acid/chondroitin sulfate
  Interventions: Drug: Hyaluronic acid/chondroitin sulfate
- Transurethral resection of bladder ulcer (Active Comparator): Transurethral resection of bladder ulcer
  Interventions: Drug: Hyaluronic acid/chondroitin sulfate

INTERVENTIONS:
Drug: Hyaluronic acid/chondroitin sulfate — Additional Hyaluronic acid/chondroitin sulfate instillation to the bladder
  Other Names: Ialuril

SUMMARY:
The purpose of this study is to evaluate efficacy and safety of additional hyaluronic acid/chondroitin sulfate to transurethral resection of bladder ulcer in patient with interstitial cystitis.

DETAILED DESCRIPTION:
This is a randomized, parallel, 6 month period study.

ELIGIBILITY:
Inclusion Criteria:

1. must have experienced bladder pain, urinary urgency and urinary frequency, for at least 6 months prior to entry into the study
2. Pain VAS ≥4
3. O'Leary-Sant Interstitial Cystitis questionnaire (IC-Q) symptom and problem ≥ 12( and pain ≥2, and nocturia ≥ 2)
4. PUF score ≥ 13
5. cystoscopic record within 2 years
6. Hunner ulcer lesion in cystoscopic finding

Exclusion Criteria:

1. Scheduled for or use of intravesical therapy (eg, bladder distention,transurethral resection of bladder ulcer, instillation) during or within 6months prior to the study and use of pentosan polysulfate sodium within 1 months prior to the study
2. Patients who are pregnancy or, childbearing age without no contraception
3. Patients with voided volume <40 or, > 400ml
4. Patients with microscopic hematuria, (≥1+ in dipstick), If not excluded that no evidence of neoplastic tumor examination
5. Patients with urine culture showing evidence of urinary tract infection 1month prior to the study
6. Accompanied medical problem below

   * Tuberculosis in urinary system
   * Bladder cancer, urethral cancer, prostate cancer
   * Recurrent cystitis
   * anatomical disorder
7. Patients had prior surgery (eq, bladder augmentation, cystectomy
8. Patients with neurologic disorder
9. Patients with indwelling catheter or intermittent self-catheterization
10. Patients with psychologic problem

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-03-20 (Actual); Primary Completion 2016-12-01 (Actual); Study Completion 2016-12-01 (Actual)

PRIMARY OUTCOMES:
Change of pain scores on the Visual Analogue Scale | 1month, 3month, 6month
  Change of pain scores on the Visual Analogue Scale

SECONDARY OUTCOMES:
Duration of symptom improvement | 1month, 3month, 6month
  Duration of symptom improvement
Changes of frequency and urgency on voiding diary | 1month, 3month, 6month
  Changes of frequency and urgency on voiding diary
Change score of O'Leary-Sant Interstitial Cystitis questionnaire (IC-Q) | 1month, 6month
  Change score of O'Leary-Sant Interstitial Cystitis questionnaire (IC-Q)
Score of Global Response Assessment (GRA), Patient Global Assessment (PGA) score | 6month
  Score of Global Response Assessment (GRA), Patient Global Assessment
Occurrence of adverse event | 6month
  Occurrence of adverse event
Change score of Pelvic Pain and Urgency/Frequency Patient Symptom Scale(PUF) | 1month, 6month
  Change score of Pelvic Pain and Urgency/Frequency Patient Symptom Scale
Change score of EQ-5D Health Questionnaire | 1month, 6month
  Change score of EQ-5D Health Questionnaire
Change score of Brief Pain Inventory-short form (BPI-sf) | 1month, 6month
  Change score of Brief Pain Inventory-short form (BPI-sf)

CONTACTS AND LOCATIONS:
Overall Officials: Myung -Soo Choo, profesor, Principal Investigator — Asan Medical Center
Locations (1):
- Asan medical center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No